CLINICAL TRIAL: NCT00536536
Title: Evaluating the Transferability of a Successful, Hospital-based, Childhood Obesity Clinic to Primary Care: a Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bristol (Other)
Responsible Party: Principal Investigator, Julian Hamilton-Shield, Professor of Diabetes and metabolic Endocrinology, University of Bristol
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PB-PG-0706-10090
Record Dates: First submitted 2007-09-27; First posted 2007-09-28 (Estimated); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Childhood Obesity
Keywords: Childhood; Obesity; Primary Care
MeSH Terms: conditions — Pediatric Obesity; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hospital (Active Comparator): Care of Childhood Obesity Clinic (COCO)
  Interventions: Behavioral: Obesity management framework
- Primary Care (Active Comparator): Primary care clinics (x2)
  Interventions: Behavioral: Obesity management framework

INTERVENTIONS:
Behavioral: Obesity management framework — Treatment in primary care will be compared to treatment in a secondary hospital setting. Treatment in both cases will be provided by a multi-disciplinary team of: obesity or practice nurse, dietitian, exercise specialist with some input from medical team.

SUMMARY:
Obesity affects one in five children in the UK and undoubtedly causes increased ill health with rising levels of childhood and adolescent diabetes, obesity induced liver disease and increased risk of early heart disease. There are few clinics offering effective treatment for childhood obesity. However, the clinic for childhood obesity at Bristol Royal Hospital for Children (BCH) has been successful in around 83% of cases. This pilot study aims to examine the feasibility of transferring the success of the hospital clinic to primary care in preparation for a full RCT. The study will entail training a practice nurse, community dietician and exercise specialist to deliver the same clinical service in primary care as that offered in BCH. Initial work will gather the views of staff delivering the hospital service and those of patients and parents to identify the crucial components of the intervention that are likely to be needed in primary care and to then to refine the intervention.A pilot trial will examine how feasible it is to recruit patients into the service and get some initial idea as to whether weight management is equally good, patient satisfaction and retention improves and what data needs to be collected for a full economic assessment. If found to be effective, the next step will be to use knowledge gained in this study to design and undertake a more extensive, formal study across Bristol in various primary care settings.This larger study will address how such a service can be delivered across a complete spectrum of primary care populations, so that similar services could be developed across the country.

DETAILED DESCRIPTION:
The care of childhood obesity clinic (COCO) at Bristol Royal Hospital for Children (BCH) provides a proven and effective treatment service for childhood obesity and is one of only a few specialist centres in the UK. The clinic service is based around a multidisciplanary team comprising: consultant; specialist nurses; dietitian: exercise specialist. This pilot study examines the feasibility of transferring the hospital clinic to a nurse led primary care setting in preparation for a full RCT. The study involves training a practice nurse to deliver the service in primary care alongside a dietitian and exercise specialist. Initial work will collect the views of staff delivering the hospital service and patients and parents which will enable us to identify the components of the service that will be needed to run a primary care based service. As a pilot we will focus on: (a) whether weight management is equally good in primary care; (b) whether recruitment, patient retention and satisfaction can be improved in primary care and (c) what data need to be collected for a full economic assessment.

Children will be recruited to the trial by GP via electronic referral form designed by the study team. Families of children fulfilling recruitment criteria (age: 5-16, BMI≥98th centile) will be sent a study pack and reply form, all those who do not respond will be contacted by the COCO consultant to clarify willingness to participate. Families declining participation will follow usual care pathway. Recruited families will be randomised to one of two primary care clinics or COCO clinic.

ELIGIBILITY:
Inclusion Criteria:

* 5 to <18 yrs old on day of recruitment
* Children consulting their general practitioner or other primary care professional with a weight > 95th percentile

Exclusion Criteria:

* Suspected underlying pathology or syndrome on primary consultation
* Severe learning difficulties

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 106 (Actual)
Dates: Start 2008-04; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
To investigate the feasibility of replicating a successful hospital based, childhood obesity clinic in primary care using trained primary care staff and undertake a pilot trial. | 12 months
  To measure whether attendance and retention are similar in primary care clinic to hospital based clinic.

SECONDARY OUTCOMES:
Primary care staff training | 12 months
  Can we train primary care staff to deliver the weight management intervention
General practice engagement | 12 months
  Is it possible to engage general practices in structured care of obese children
Family expectations of locality based, weight management clinics. | 12 months
  What parents and children would like to see in a community based service especially regarding access and retention in the service
Defining outcomes for main RCT. | 12 months
  The optimum outcome measures to be used in the main RCT especially for the health economics
The protocol for GP screening to identify exclusions | 3 months
  To produce a GP exclusion criteria list for main RCT.
Sample size calculation (for main trial) | 24 months
  The likely size of differences between the groups and thus the size of the main trial

CONTACTS AND LOCATIONS:
Overall Officials: Debbie Sharp, Principal Investigator — University of Bristol; Christopher Salisbury, Principal Investigator — University of Bristol
Locations (1):
- Bristol Primary Care Trust, Bristol, United Kingdom

REFERENCES:
- [Derived] Hollinghurst S, Hunt LP, Banks J, Sharp DJ, Shield JP. Cost and effectiveness of treatment options for childhood obesity. Pediatr Obes. 2014 Feb;9(1):e26-34. doi: 10.1111/j.2047-6310.2013.00150.x. Epub 2013 Mar 18. PMID 23505002
- [Derived] Banks J, Sharp DJ, Hunt LP, Shield JP. Evaluating the transferability of a hospital-based childhood obesity clinic to primary care: a randomised controlled trial. Br J Gen Pract. 2012 Jan;62(594):e6-12. doi: 10.3399/bjgp12X616319. PMID 22520658
- [Derived] Banks J, Williams J, Cumberlidge T, Cimonetti T, Sharp DJ, Shield JP. Is healthy eating for obese children necessarily more costly for families? Br J Gen Pract. 2012 Jan;62(594):e1-5. doi: 10.3399/bjgp12X616300. PMID 22520655